CLINICAL TRIAL: NCT06223568
Title: Phase II Trial of Neoadjuvant Chemotherapy (NAC) Alone or in Combination With Immunotherapy Vaccine PRGN-2009 in Subjects With Newly Diagnosed HPV-Associated Oropharyngeal (Head and Neck) Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001730; 001730-C
Record Dates: First submitted 2024-01-24; First posted 2024-01-25 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-14

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Oropharynx; Human Papillomavirus Viruses; Drug Therapy; Cancer Vaccine
Keywords: Neoadjuvant Chemotherapy; Oropharynx Cancer; Human Papillomavirus; Therapeutic Vaccine
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): DC (docetaxel + cisplatin)
  Interventions: Drug: Docetaxel; Drug: Cisplatin
- Arm 2 (Experimental): DCP (docetaxel + cisplatin + PRGN-2009)
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: PRGN-2009

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m^2 will be administered over 60 (+/-10) minutes.
Drug: Cisplatin — Cisplatin 75 mg/m^2 will be administered over 120 (+/-10) minutes.
Drug: PRGN-2009 — PRGN-2009 will be administered in Arm 2 participants only as an SQ injection in the arm at a dose of 1 mL nominally containing 5x10^11 viral particles (VP) on Day -7 (+/-3 days) of Cycle 1, Day 11 (+/-3 days) of Cycles 1, 2, and 3.
  Arms: Arm 2

SUMMARY:
Background:

Throat cancer is a common tumor that can occur in people infected with the human papilloma virus (HPV). Most people with this cancer survive more than 5 years with standard chemotherapy drugs plus radiation. But radiation can cause serious adverse effects. Researchers believe that adding a vaccine (PRGN-2009) to this drug therapy may improve survival without the need for radiation.

Objective:

To test a study vaccine combined with standard chemotherapy in patients with HPV-associated throat cancers.

Eligibility:

People aged 18 years and older with newly diagnosed throat cancer associated with HPV.

Design:

Participants will be screened. They will have a physical exam and blood tests. They will have imaging scans and tests of their heart function and hearing. They will provide a sample of tissue from their tumor. A recent sample may be used; if none is available, a new sample will be taken.

All participants will get two common drugs for treating cancer. These drugs are given through a tube attached to a needle inserted into a vein in the arm. Participants will receive these drugs on the first day of three 3-week cycles.

Half of the participants will also get the vaccine. PRGN-2009 is injected under the skin in the arm. They will get these shots 4 times: 7 days before the start of the first cycle and on the 11th day of each cycle.

Participants will have standard surgery to remove their tumors 3 to 6 weeks after completing the study treatment. They will have follow-up visits 3, 6, 12, and 24 months after their surgery.

...

DETAILED DESCRIPTION:
Background:

* Human papilloma virus (HPV)-associated oropharyngeal squamous cell carcinoma (OPSCC) is among the most common HPV-associated malignancies and the incidence is increasing. The prognosis is favorable with >80% 5-year recurrence free survival observed following standard anti-cancer treatments that consist of surgery followed by adjuvant post-operative radiation therapy (PORT) or concurrent chemoradiation (CRT).
* Although oncologic control is excellent, these standard-of-care treatments often lead to radiation-associated long-term toxicity that includes tissue fibrosis resulting in long-term swallow dysfunction and poor quality of life (QOL).
* Neoadjuvant chemotherapy (NAC) followed by surgery has decades of real-world data, with clinical-to-pathologic downstaging or pathologic complete response (pCR) being observed in most patients, >90% 5-year survival, and complete avoidance of radiation treatment in >95% of patients.
* The rate of pCR, clinical-to-pathologic downstaging, and functional outcomes after NAC followed by surgery have not been studied in a formal, prospective clinical study.
* A pilot correlative study of NAC with docetaxel and cisplatin (DC) in patients with newly diagnosed HPV-associated OPSCC conducted at the NIH revealed induction of HPV-specific T cell immunity that associates with clinical outcome (18DC0051).
* PRGN-2009 is a gorilla adenoviral therapeutic vaccine designed to enhance HPV 16/18- specific T-cell responses. The safety and efficacy of PRGN-2009 in patients with newly diagnosed HPV-associated OPSCC have been studied at the NIH Clinical Center (NCT04432597).
* Pre-clinical data indicate that chemotherapy can remodel the tumor microenvironment and enhance immunotherapy, suggesting that the combination of DC and PRGN-2009 may enhance anti-tumor immunity and the rate of pCR beyond that observed with DC alone.

Objective:

-To determine the rate of pCR with NAC (DC) alone or in combination with PRGN-2009 (DCP) in participants with newly diagnosed HPV-associated OPSCC.

Eligibility criteria:

* Pathologically confirmed newly diagnosed surgically resectable stage I or II HPV-positive oropharyngeal squamous cell carcinoma.
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2 and adequate organ function.

Design:

* Participants diagnosed in the community with newly diagnosed HPV-associated OPSCC will be referred to the NIH Clinical Center for neoadjuvant treatment.
* Participants will be randomized to receive either DC (Arm 1) or DCP (Arm 2) in the neoadjuvant setting. DC is three cycles of intravenous cisplatin plus docetaxel, administered every 21 days. PRGN-2009 is 4 doses of subcutaneous vaccination administered on Day -7 of Cycle 1, and Day 11 of Cycles 1, 2, and 3. Participants will be stratified at registration for stage (I or II).
* Participants will undergo pre- and post-treatment Positron Emission Tomography (PET) / Computed Tomography (CT) and measurement of circulating cell-free HPV DNA.
* Participants will return to the community to receive standard-of-care surgery. The need for pathology-indicated, risk-stratified PORT will be determined per standard of care.
* Pathologic responses and follow-up to assess swallow function, QOL, hearing function, and recurrence-free survival will take place at the NIH Clinical Center.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed surgically resectable newly diagnosed stage I (cT1-2, N0-1) or II (T1-3, N0-2), M0 oropharyngeal squamous cell carcinoma. Note: Pathological report of cancer diagnosis may be from the primary tumor or from a metastatic cervical lymph node.
* History of HPV-positive status determined by a standard-of-care HPV testing. Note: All participants with high-risk HPV serotypes are eligible.
* Age >= 18 years.
* ECOG performance status <= 2.
* Individuals who smoke currently must smoke <10 pack years. Note: Former smokers with any pack-year history are eligible if quit smoking >10 years before study treatment initiation. Former smokers who quit <10 years before study treatment initiation must have smoked <10 pack years.
* Planned for cancer removal surgery per standard of care (SOC) and individual had agreed for the cancer removal surgery.

  * Individuals must have adequate organ and marrow function as defined below:
  * Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
  * Hemoglobin (Hgb) >= 9.0 g/dL
  * Platelet count >= 100 x 10^9/L
  * Creatinine <= 1.2 x upper limit of normal (ULN) OR calculated creatinine clearance >=55 mL/min/1.73m^2 by Cockcroft-Gault formula
* Total bilirubin <= 1 x ULN, or <= 3 x ULN in patients with known or suspected Gilbert's Syndrome
* Alanine aminotransferase (ALT) <= 1.5 x ULN
* Aspartate aminotransferase (AST) <= 1.5 x ULN
* Individuals serologically positive for human immunodeficiency virus (HIV) must:

  * be on effective anti-retroviral therapy for at least 4 weeks; and
  * have undetectable viral load; and
  * have the CD4 count >=200 cells/microL; and
  * have no reported opportunistic infections or Castleman s disease within 12 months prior to study treatment initiation
* Individuals serologically positive for Hepatitis C virus (HCV) or Hepatitis B virus (HCB) must have an undetectable viral load.
* Individuals of child-bearing potential (IOCBP) must agree to use a highly effective method of contraception (hormonal, intrauterine device (IUD), surgical sterilization, abstinence) for the duration of the study treatment and up to 2 months after the last dose of PRGN-2009 and an effective method of contraception (barrier, hormonal, intrauterine device (IUD), surgical sterilization, abstinence) for 14 months after the last dose of cisplatin/docetaxel. Note: IOCBP is defined as any woman who has experienced menarche and has not had a hysterectomy or bilateral oophorectomy or is not postmenopausal (amenorrheic 12 months or more following cessation of exogenous hormonal treatments; if <50 years old and need follicle stimulating hormone [FSH] in the post-menopausal range).

Men must agree to use a highly effective method of contraception (surgical sterilization, abstinence) for the duration of the study treatment and up to 2 months after the last dose of PRGN-2009 and an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and up to 11 months after the last dose of the study drug(s). We also will recommend men on treatment with PRGN-2009 with female partners of childbearing potential ask female partners to be on highly effective birth control (hormonal, intrauterine device (IUD), surgical sterilization) during PRGN-2009 treatment and 2 months after that.

* Breastfeeding individuals must be willing to discontinue breastfeeding from study treatment initiation through 2 months after the last dose of the study drug(s).
* Individuals must have a tumor site that is amenable to biopsy and be willing to undergo pre- treatment biopsy for research purposes.
* Individuals must be willing to undergo pre-treatment PET/CT imaging study.
* The ability of an individual to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Peripheral motor or sensory neuropathy > Grade 2 per Common Terminology Criteria for Adverse Events (CTCAE) v.5 at screening.
* Prior therapy with an investigational drug, live vaccine, chemotherapy, immunotherapy, or any prior radiotherapy (except for palliative bone-directed therapy) within 4 weeks prior to the first study drug administration. Note: Participants may continue adjuvant hormonal therapy in the setting of a definitively treated cancer (e.g., breast).
* Prior therapy with any medications or substances that are moderate or strong inducers or moderate or strong inhibitors of cytochrome P450 (CYP3A) https://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm#table2-2,table3-3,table5-2 within 2 weeks prior to the first study drug administration.
* History of allergic reactions attributed to compounds of similar chemical or biological composition to drugs used in the study.
* Systemic (intravenous or oral) glucocorticoid (except for physiologic doses of corticosteroids, i.e., <= the equivalent of prednisone 10 mg/day) or other immunosuppressors such as azathioprine or cyclosporin A within 1 week prior to study treatment initiation. Note: Glucocorticoids as premedication for contrast-enhanced studies are allowed.
* Second malignancy active within the previous 2 years except for indolent or locally curable malignancy that is currently considered cured and/or does not require an additional standard of care treatment, such as, but not limited to, cutaneous basal or squamous cell carcinoma, superficial bladder cancer, or cervical carcinoma in situ, or an incidental histological finding of prostate cancer or differentiated thyroid cancer.
* Prior allogenic tissue/solid organ transplant.
* History of heart failure.
* Positive beta-human chorionic gonadotropin (beta-HCG) serum or urine pregnancy test performed in females of childbearing potential at screening.
* Uncontrolled intercurrent illness or medical condition(s) evaluated by medical history and physical exam or situations that are not stable (e.g., recent hospitalization, Emergency Room visit or undergoing medication changes) that would potentially increase risk for the participant.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2028-01-10 (Estimated); Study Completion 2028-01-10 (Estimated)

PRIMARY OUTCOMES:
Determine the rate of pCR with NAC (DC) alone or in combination with PRGN-2009 (DCP) in participants with newly diagnosed HPV-associated OPSCC | 6 months
  The pCR rates will be determined on each arm and will be reported along with a 95% confidence interval. The two rates will be compared using a one-sided Fisher s exact test.

SECONDARY OUTCOMES:
Determine the toxicity observed with DC and DCP | Day 1 (all arms) and day 11 (Arm 2 only) of every cycle and Day -7 of C1 (Arm 2 only), and at Safety Follow-Up visit which occurs 14 (+14) days after the study agent (s) was/were last administered. 3-month follow-up visit and beyond.
  Safety will be evaluated by determining the frequency of adverse events among treated participants and reporting the results, by maximum grade of event and type of toxicity noted. Tolerability will be recorded in the form of number of participants that discontinued treatment, had a delay in any study treatment or a DC dose reduction, and any study drug-related surgical delays.
Determine 2-year recurrence-free survival (RFS) observed with DC and DCP | 3, 6, 12, 24 months after surgery per SOC until recurrence.
  Recurrence-free survival will be determined using the Kaplan-Meier method for each arm, with recurrence or death without recurrence considered as events. The two-year recurrence-free survival values will be reported along with a 95% two-sided confidence interval for each arm. The two curves will also be compared using a two-tailed log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Clint T Allen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001730-C.html